CLINICAL TRIAL: NCT00897039
Title: Application of the Microculture Kinetic (MiCK) Assay for Apoptosis to Testing Drug Sensitivity of Ovarian, Fallopian and Primary Peritoneal Adenocarcinomas
Brief Title: Laboratory Study in Predicting Tumor Response to Chemotherapy in Patients With Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeastern Gynecologic Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000491440; SEG-20060042; SEG-IRB-1075624
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-07

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: ovarian serous cystadenocarcinoma; ovarian undifferentiated adenocarcinoma; recurrent ovarian epithelial cancer; ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian mucinous cystadenocarcinoma; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; recurrent primary peritoneal cavity cancer; stage IA primary peritoneal cavity cancer; stage IB primary peritoneal cavity cancer; stage IC primary peritoneal cavity cancer; stage IIA primary peritoneal cavity cancer; stage IIB primary peritoneal cavity cancer; stage IIC primary peritoneal cavity cancer; stage IIIA primary peritoneal cavity cancer; stage IIIB primary peritoneal cavity cancer; stage IIIC primary peritoneal cavity cancer; recurrent fallopian tube cancer; stage IA fallopian tube cancer; stage IB fallopian tube cancer; stage IC fallopian tube cancer; stage IIA fallopian tube cancer; stage IIB fallopian tube cancer; stage IIC fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Flow Cytometry; Immunohistochemistry

INTERVENTIONS:
Other: flow cytometry
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: Collecting samples of tissue from patients with cancer to study in the laboratory may help doctors predict how well patients will respond to treatment with certain chemotherapy drugs and plan the best treatment.

PURPOSE: This laboratory study is looking at tumor tissue samples to predict response to chemotherapy in patients with ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the ability of the microculture kinetic (MiCK) assay to predict the outcome of patients with ovarian, fallopian tube, or primary peritoneal adenocarcinoma treated with first-line chemotherapy.
* Evaluate the ability of the MiCK assay to guide chemotherapy in a third-line, refractory treatment setting (exclusive of anti-vascular endothelial growth factor) in these patients.

OUTLINE: Patients are stratified according to prior chemotherapy (no [stratum I] vs yes [stratum II]).

Tumor tissue and/or effusion specimens are collected at baseline. Specimens are examined by the microculture kinetic (MiCK) assay and immunocytochemical or flow cytometry assay.

MiCK assay results do not influence treatment for stratum I patients. Stratum II patients may receive treatment based on MiCK assay results for tumor sensitivity to specific chemotherapy drugs.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed adenocarcinoma of 1 of the following types:

  * Ovarian
  * Primary peritoneal
  * Fallopian tube
* Must meet 1 of the following criteria:

  * De novo malignancy with no prior chemotherapy
  * Advanced refractory malignancy with ≤ 2 standard chemotherapy treatment protocols
* Tumor must be accessible for biopsy or drainage of effusions
* Chemotherapy is considered a treatment option
* No symptomatic or uncontrolled parenchymal brain metastases
* No meningeal metastasis

PATIENT CHARACTERISTICS:

* Not pregnant
* Negative pregnancy test
* Fertile patients must agree to use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Correlation of a statistically significant discriminator of sensitivity with complete response rate

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir D. Kravtsov, MD, Study Chair — Pierian Biosciences; Matthew O. Burrell, MD — Southeastern Gynecologic Oncology
Locations (1):
- Southeastern Gynecologic Oncology, LLP - Northside, Atlanta, Georgia, United States